# Intra-operative Steroid Irrigation for Reducing Recurrent Laryngeal Nerve Palsy Post-thyroidectomy – A Pilot Study

Study Duration: 1/11/2024 - 31/10/2026

# Kah Seng Khoo<sup>a</sup>

MBBS (UM)

MRCS (Edinburgh)
MSurg (UM)

## Joanne Aisha Mosiun<sup>a</sup>

MBBS(UM)

MRCS (Edinburgh)

MSurg (UM)

## Redzwan Shah Bin John Mohd<sup>b</sup>

MBBS (UM), MSORLHNS (UM)

#### Yoke Kiet Doon<sup>a</sup>

MD (MOSCOW)

MSurg (UM)

# Khoon Leong Ng<sup>a</sup>

MBBS (S'pore)

FRCS (Glasg) FRCS (Ed)

AM (Mal)

# Mee Hoong See<sup>a</sup>

MD (UPM)

MSurg (UM)

a Breast & Endocrine Surgery Unit, Department of Surgery, University of Malaya, Malaysia

b Department of Otorhinolaryngology, University of Malaya, Malaysia

\*Corresponding author: Kah Seng Khoo, Tel: +6017-2489272, Email: kahseng901209@gmail.com

Date of document: 1/11/2024



#### **Patient Consent Form**

| Name: |
|-------------------|
| Date of Birth: |
| IC Number: |
| Address: |
| Telephone Number: |

I consent to participate in the above research study.

I understand that if I agree to participate, I also agree to disclose my medical history. I authorize members of the research team to have access to and view my pathology report and medical records.

I understand that information obtained during this study will be securely stored on an electronic database and will not be used for any other purposes. I also understand that my participation in this study is entirely voluntary and that I may withdraw from any or all parts of it, at any time, without giving a reason and without affecting my further care.

| ••••• | ••••• | ••••• |
|---------------------|--------------------------|-------|
| Name of Participant | Signature of Participant | Date |
| | | ••••• |
| Name of Person | Signature | Date |
| Obtaining Consent | | |